CLINICAL TRIAL: NCT06315114
Title: A Transdiagnostic Mentalization-based Intervention (LIGHTHOUSE Parenting Program) Versus Care as Usual for Parents With Mental Disorders in Adult Mental Health Service: a Randomised Clinical Trial
Brief Title: A Transdiagnostic Mentalization-based Intervention for Parents With Mental Disorders
Acronym: LIGHTHOUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p-2023-15049; H-23064491 (Other: Regional Committee of Health Research Ethics (VEK))
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Mental Disorder; Behavior Disorders; Diagnosis, Psychiatric; Diagnosis Dual; Severe Mental Disorder; Mental Illness; Psychiatric Disorder; Psychiatric Disease; Psychiatric Illness
Keywords: Mental disorder; Parent; Child; Preventive intervention; Prevention; Intergenerational transmission
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lighthouse MBT Parenting Program (LPP) (Experimental): The experimental group is a manualized transdiagnostic mentalization-based parenting intervention (Lighthouse MBT Parenting Program). This is a 12-week parenting group intervention (weekly session of 2 hours) with one preperatory initial individual session (1 hour) before the group commence.
  Interventions: Behavioral: Lighthouse MBT Parenting Program (LPP)
- Care as usual (CAU) (Active Comparator): 1-2 next of kin sessions (called 'Familiesamtale') is considered the care as usual offered to parents in adult mental health service in the Capital Region of Denmark.
  Interventions: Behavioral: Care as usual (CAU)

INTERVENTIONS:
Behavioral: Lighthouse MBT Parenting Program (LPP) — The experimental group is a manualized transdiagnostic mentalization-based parenting intervention (Lighthouse MBT Parenting Program). This is a 12-week parenting group intervention (weekly session of 2 hours) with one preperatory initial individual session (1 hour) before the group commence.
  Arms: Lighthouse MBT Parenting Program (LPP)
Behavioral: Care as usual (CAU) — 1-2 next of kin sessions (called 'Familiesamtale') is considered the care as usual offered to parents in adult mental health service in the Capital Region of Denmark.
  Parents are offered the possibility of bringing their spouse or offspring to one of the sessions.
  Arms: Care as usual (CAU)

SUMMARY:
The aim of this randomised clinical trial is to evaluate the short and longterm effects of a transdiagnostic mentalization-based intervention (Lighthouse MBT Parenting Program) compared to care as usal (CAU) for parents with a mental disorder in adult mental health service.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), 970 million people worldwide suffer from mental disorders, many of whom are parents. Cross-sectional studies indicate that between 15-55% of the patients attending adult mental health service (AMHS) are parents. In Denmark, about 430.000 children have at least one parent with a mental disorder.

Parental mental health problems have a detrimental impact on parenting, leading to long-term negative consequences for their children. Robust evidence shows that children of parents with mental disorders have an elevated risk of various adverse outcomes and events, such as developing a mental disorder themselves and exposure to child maltreatment, compared to children of healthy unaffected parents, suggesting an intergenerational transmission of adversity from parent to child. Mental disorders in parents thus leaves deep traces throughout their children's' lives and entails major socio-economic consequences. Given the high prevalence and substantial burden of parental mental disorders, there is an urgent need for evidence-based interventions targeting the specific needs of this population to prevent the adverse impact on their children. Despite this, the existing services in AMHS for parents with mental disorders are insufficient, and not evidence based. The present trial seeks to fill in this gap.

This is an investigator-initiated single-center, two-arm, parallel group randomized clinical trial testing for superiority of a transdiagnostic mentalization-based intervention (Lighthouse MBT Parenting Program) versus care as usual in 170 parents with various mental disorders. The experimental intervention and active control group intervention are delivered as an add-on to the participants' outpatient treatment.

Participants will be recruited from the outpatient clinics at Psychotherapy Centre Stolpegaard (PCS), Capital Region of Denmark. Participants will be included if they comply with the eligibility criteria. Participants will be assessed at baseline, and at 6, 12, and 24 months follow-up after randomization.

ELIGIBILITY:
Inclusion Criteria exclusive to the Outpatient Clinic

* Age >18 years
* Seeking treatment for one of the following non-psychotic disorders according to ICD-10: obsessive-compulsive disorder and anxiety disorders (F40-42), posttraumatic stress disorder (DF43), personality disorders (F60-61), or one of the previous disorders and a drug-or alcohol related disorder (F10-19) (i.e. 'dual diagnosis disorder')

Inclusion Criteria exclusive to the trial:

* Parent of at least one child aged 0-17 years of age at baseline
* Fluent i.e., sufficient Danish language skills
* Parent is living with child or is in regular contact (min. 5 days monthly)
* Written informed consent

Exclusion Criteria exclusive to the Outpatient Clinic:

* Possibility of a learning disability (IQ<75)
* A diagnosis of schizotypal personality disorder or antisocial personality disorder
* Presence of a comorbid psychiatric disorder that requires specialist treatment elsewhere
* Concurrent psychotherapeutic treatment outside the clinic

Exclusion Criteria exclusive to the trial:

* Acute suicidal risk or state of crises
* Lack of informed consent
* Acute child endangerment
* Participation in another parenting focused intervention simultaniously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Parenting stress assessed with Parenting Stress Index - Short Form (PSI-4-SF) | Baseline, and at 6, 12, and 24 months post randomization
  PSI-4-SF is a 36-item questionnaire assessing self-reported levels of parenting stress. The PSI-4-SF consists of three subscales: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC). A total stress score indicates the overall level of parenting stress as experienced by the parent. Parents rate the degree to which they agree with each statement (SA: Strongly agree, A: Agree, NS: Not sure; D: Disagree, SD: Strongly Disagree). Range: 36-180 with higher scores indicating higher levels of parenting stress.

SECONDARY OUTCOMES:
Psychological adjustment in children assessed with the Strenght and Difficulties Questionnaire - Extended version (SDQ) | Baseline, and at 6, 12, and 24 months post randomization
  SDQ is a 25-item questionnaire assessing parent-reported child emotional and behavioural problems. The SDQ has five scales (scored 0-10); emotional problems, conduct problems, hyperactivity, peer problems and pro-social scale. The scales are combined (excluding the pro-social scale) into a 'total difficulties' score (Range: 0-40, with higher scores indicating more problems). The items on the overall distress and impairment can be summed to generate an impact score (Range: 0-10), indicating the need for assessment and possible intervention. Parents rate the degree to which they agree with each statement (NT: Not true, ST: Somewhat true, CT: Certainly true). Higher scores indicate more problems or more functional impairment.
Quality of life in parents assessed with the World Health Organization Questionnaire of Life - BREF (WHOQL-BREF) | Baseline, and at 6, 12, and 24 months post randomization
  WHOQL-BREF is a 26-item questionnaire assessing self-reported quality of life. The instrument measures an individual's overall quality of life and general health and four health dimensions: Physical health, psychological, social relationships, and environment. The domain scores are scaled in a positive direction with higher scores indicating a higher quality of life. The two domains assessing psychological health (6 items) and social relationsships (3-items) and the measure of the overall quality of life and general health (2 items) will be used.
Family functioning assessed with the McMaster Family Assessment Device - General Functioning Scale (FAD-GF). | Baseline, and at 6, 12, and 24 months post randomization
  The FAD is a questionnaire assessing self-reported perceptions of the parent's current family relationships. It consists of five subscales: problem solving, communication, roles, affective responsiveness, affective involvement, behavior control, and general functioning. Parents rate each statement on a 4-point scale (SA: Strongly agree, A: Agree, D: Disagree, SD: Strongly Disagree). Only the general functioning (6-items) subscale will be used.Range: 6-24, with higher scores indicating more functional impairment.
Childhood adversity in children assessed with the Adverse Child Experciences Questionnaire (ACE) extended version developed by the Center for Youth Wellness (CYW) | Baseline, and at 6, 12, and 24 months post randomization
  ACE CYW is questionnaire assessing parent-reported childhood adversity in children and adolescents. The instrument is comprised of two sections: Section 1 consists of the traditional ten ACEs covering exposure to childhood psychological, physical, and sexual abuse as well as household dysfunction, including domestic violence, substance use, and incarceration. Section 2 includes seven (CYW ACE-Q Child) or nine (CYW ACE-Q Teen) items assessing for exposure to additional early life stressors, including involvement in the Foster Care system, bullying, loss of parent or guardian due to death, deportation or migration, medical trauma, exposure to community violence, and discrimination. Parents are asked to how many categories apply to their child (i.e. they do not specificy which categories applies). Parents tally the number for each section, and report the total number, thus resulting in two total scores. Higher scores indicates exposure to more adverse events.
Parenting competence assessed with the Parenting Sense of Competence (PSOC) | Baseline, and at 6, 12, and 24 months post randomization
  PSOC is a 16-item questionnaire assessing self-reported parenting competence It consists of 2 subscales: Parental satisfaction and parental self-efficacy. Parents rate each item on a 6-point scale.ossible scores range from 10 to 60 for Efficacy and 6 to 36 for Satisfaction. Lower scores may indicate a parent's uncertainty about whether they have the knowledge or skills required to be an effective parent.
Psychiatric symptom severity in parents assessed with the Brief Symptom Inventory (BSI) | Baseline, and at 6, 12, and 24 months post randomization
  BSI is a 53-item questionnaire assessing self-reported severity of psychiatric symptoms adapted from the Symptom Checlist Revised (SCL-90-R). it covers 9 symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. The global indices measure current or past level of symptomatology, intensity of symptoms, and number of reported symptoms, respectively. Parents rate each statement on a 5-point scale ranging from 0 (not at all ) to 4 (extremely). Range: 0-212, with higher scores indicating higher symptom severity
Health related quality of life and functioning in parents assessed with the European Quality of life - 5 Dimensions (EQ-5D) | Baseline, and at 6, 12, and 24 months post randomization
  EQ-5D is a 5-item questionnaire assessing health related quality of life and level of functioning. Parents select one out of three statements within each of five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Higher scores indicates better quality of life. The statements are complemented by a visual analog scale in which parents are asked to rate the health ranging form 0 (worst imaginable health) to 100 (best imaginale health)

OTHER OUTCOMES:
Parental mentalizing assessed with the Parental Reflective Functioning Questionnaire (PRFQ) | Baseline, and at 6, 12, and 24 months post randomization
  PRFQ is a 18-item questionnaire assessing self-reported parental mentalizing.Higher scores on the PM indicates impaired mentalizing, while high and low scores on IC and CMS indicates impaired mentalizing.
Mind-mindedness assessed with the Representational Mind-Mindedness (MM) interview | Baseline and at 6 months post randomization
  In the MM interview, parents are asked to describe their child. The response is taped and verbatim transcribed. The description is the coded following the guidelines from the coding manual (Meins & Fernyhough, 2015). Total score range: 0-150, with higher scores indicating better mentalizing.
Epistemic trust assessed with the Epistemic Trust, Mistrust, and Credulity Ques-tionnaire (ETMCQ) | Baseline and at 6 months post randomization
  ETMCQ is a 18-item questionnaire assessing self-reported trust in others. Higher scores on trust indicates higher levels of trust, while higher scores on mistrust and credulity indicates epistemic mistrust.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Simonsen, Doctor, Study Director — Mental Health Service, Capital Region, Denmark
Locations (2):
- Denmark (2):
  - Psychotherapeutic Centre Stolpegaard, Gentofte Municipality, Capital Region
  - Psychotherapeutic Centre Stolpegård, Gentofte Municipality

IPD SHARING:
Plan to Share IPD: Yes
No plan yet
Supporting Information: Study Protocol, ICF
Time Frame: Fall 2028
Access Criteria: For more information contact PI

REFERENCES:
- See also: Profile of project leader — http://www.researchgate.net/profile/Emilie-Hestbaek-2/publications
- See also: Description of trial — http://www.psykiatri-regionh.dk/fagfolk/forskning-i--region-hovedstadens-psykiatri/forskningsomraader/Udvalgte%20projekter/Sider/LIGHTHOUSE-projektet.aspx